CLINICAL TRIAL: NCT05793931
Title: Breaking Down Financial Barriers: A Pilot Study to Determine the Feasibility, Acceptance, and Effectiveness of In-vitro Maturation in Patients Without IVF Coverage
Brief Title: A Pilot Study to Determine the Feasibility, Acceptance, and Effectiveness of In-vitro Maturation in Patients Without IVF Coverage
Acronym: IVM
Status: Terminated | Type: Observational
Why Stopped: Funding expired 03/01/2023
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: STU00213583
Record Dates: First submitted 2023-02-21; First posted 2023-03-31 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: IVM; PCOS
Keywords: IVM; PCOS; PCAO

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specific aim of this pilot study is to test the hypothesis that estrogen stimulated IVM will be non-inferior to traditional IVF, to determine the feasibility and acceptance of estrogen-stimulated in vitro maturation (IVM) among couples and if couples find value and satisfaction with IVM.

This project will determine the feasibility, acceptance, and cost-benefit of in vitro maturation (IVM) among 20 couples who have had unsuccessful attempts at pregnancy using oral medications or whose only option to achieve pregnancy is through in vitro fertilization (IVF) due to blocked fallopian tubes or low sperm counts.

DETAILED DESCRIPTION:
Initial treatment for infertility often involves the use of ovulation induction with or without intrauterine insemination. This is particularly useful in the large number of PCOS patients seeking care. However, 30-50% of couples fail such treatments and are recommended to pursue in vitro fertilization (IVF). While IVF remains the most effective of all infertility treatments, it is also the most expensive. The CDC's 2014 report on the utilization of infertility services in the U.S. estimated that between 2006-2010 approximately 67% of reproductive-aged women sought infertility services (advice, evaluation, and/or treatment). Of these women, only 6.9% used artificial insemination and 2.6% used IVF.

In addition to improving access to IVF treatment by lowering costs, IVM has the potential to make IVF treatment safer for women. The injectable medications used in IVF often overstimulate the ovaries and can lead to developing a dangerous syndrome called ovarian hyperstimulation syndrome (OHSS). OHSS is a condition in which significant fluid shifts occur within a woman's blood vessels which can lead to ascites, pulmonary edema, difficulty breathing, and in rare cases, death. OHSS also poses the risk of severe blood clotting which can lead to heart attack, stroke, and pulmonary embolism - all potential lethal complications.

In vitro maturation (IVM) is a technique where immature eggs are aspirated from the ovary without the use of injectable medications. The eggs are cultured to maturity in the laboratory which enables them to be fertilized. They are then fertilized in the laboratory and transferred back to the mother's uterus similar to traditional IVF. With improvements in IVM technique, recent data have shown that IVM can produce near comparable pregnancy rates to IVF and eliminate OHSS.

Our goal is to determine the feasibility, acceptance, and effectiveness of IVM in couples who have a female partner with PCOS or polycystic appearing ovaries (PCAO). With the cost of traditional IVF ranging anywhere from $12,000 - $15,000 per cycle, the estimated $2,500- $4,000 cost of IVM may be a more cost-effective and safer strategy among couples. The results of this study not only have the potential to improve equity among those seeking infertility treatment, but also present an opportunity to serve as a springboard for future research aimed at advancing the care of all patients who seek fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients without insurance coverage for IVF
2. Female partner between age 18-3540
3. Female partner with a diagnosis of polycystic ovarian syndrome (PCOS) or polycystic appearing ovaries (PCAO) as defined by an antral follicle count ≥ 15
4. Presence of both ovaries
5. Female partner with body mass index (BMI) of 19-4035 kg/m2
6. Female partner with a normal uterine cavity as assessed by hysteroscopy, hysterosalpingography, or sonohysterography within the last 12 months
7. Female partner with a history of tubal sterilization OR Blocked fallopian tubes without evidence of a hydrosalpinx OR History of 3 or more previously failed cycles of ovulation induction with oral medications OR where IVF is recommended for the treatment of mild or moderate male factor infertility OR evidence of a polyp and infertility
8. Male partner between age 18-45
9. Male partner must be able to produce fresh semen sample
10. Male partner with sperm concentration ≥ 5 million sperm/mL and sperm motility ≥ 25%
11. English speaking

Exclusion Criteria:

1. Frozen sperm source
2. Presence of ovarian pathology (i.e., endometrioma, fibroma)
3. History of HIV or acute hepatitis infection
4. History of chemotherapy or pelvic radiation therapy
5. Any active, uncontrolled, clinically significant medical condition as determined by the investigator
6. Contradiction to pregnancy
7. Adults unable to consent
8. Pregnant women
9. Prisoners

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We seek to recruit 20 couples that fit the inclusion criteria as stated above.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Statistical analysis of live birth rates from IVM | From treatment start to live birth (~10 months)
  Measurements for analysis include: gestational age at delivery, mode of delivery, birth weight, gender, neonatal and obstetric complications

SECONDARY OUTCOMES:
Statistical analysis of IVM on oocyte retrieval and maturation | From treatment start to day 3 or day 5 of blastocyst development (~3 weeks)
  The antral follicle count (AFC), number of eggs retrieved, number of eggs mature, number of eggs fertilized, number of eggs discarded, number of embryos transferred, number of embryos frozen will be assessed together to determine efficacy of IVM on oocyte maturation to embryo stage.
Statistical analysis of IVM on embryo parameters | From fertilization to day 3 or day 5 of blastocyst development (up to 1 week)
  The number of gestational sacs present, morphology and morphokinetic embryo parameters will be combined to report statistical analysis of embryo development from IVM.
Efficacy of IVM on pregnancy | From treatment start to birth or loss (up to 10 months)
  The rate at which IVM results in not pregnant, biochemical, clinical pregnancy, miscarriage, ectopic, or pregnancy of unknown location.
Statistical analysis of IVM on endometrial response to hormones | From treatment start to hCG trigger (~2 weeks)
  The endometrial thickness on day of hCG trigger and number of total days of estrogen prior to hCG will be combined to assess the endometrial response to estrogen.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States